CLINICAL TRIAL: NCT07388186
Title: Effectiveness of a Combined Strength Training and Progressive Muscle Relaxation Program in Reducing Frailty in Informal Caregivers of People With Alzheimer's Disease: A Randomized Controlled Trial
Brief Title: Benefits of Strength Training in Informal Caregivers of Patients With Alzheimer's Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Collaborators: Colegio Profesional de Fisioterapeutas de Castilla y León (Unknown); CRE Alzheimer del Imserso (Unknown)
Responsible Party: Principal Investigator, Andrea Calleja Caballero, Physical therapist, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STRENGTH_CAREGIVERS_ALZ
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Caregiver Burden; Anxiety
Keywords: Frailty; Strength; Caregiver; Anxiety; Burden; Alzheimer disease
MeSH Terms: conditions — Frailty; Caregiver Burden; Anxiety Disorders; Alzheimer Disease | interventions — Autogenic Training

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel intervention arms and will receive either progressive muscle relaxation alone or a combined program of functional strength training and progressive muscle relaxation over a 10-week period.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Muscle Relaxation (Active Comparator): Participants in this arm will receive one weekly session of progressive muscle relaxation over a 10-week period. Each session will last approximately 45 minutes and will include diaphragmatic breathing, Jacobson's progressive muscle relaxation technique, controlled breathing exercises, and a brief cooldown period. Sessions will be supervised by a trained physiotherapist.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Strength Training plus Progressive Muscle Relaxation (Experimental): Participants in this arm will receive a combined intervention consisting of one weekly session of progressive muscle relaxation and one weekly session of functional strength training over a 10-week period. Strength training sessions will focus on upper limb, lower limb, and core muscle groups using progressive resistance. Each session will last approximately 45 minutes and will be supervised by a trained physiotherapist.
  Interventions: Behavioral: Progressive Muscle Relaxation; Behavioral: Functional Strength Training

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — Progressive muscle relaxation will be delivered in weekly supervised sessions over a 10-week period. Each session will last approximately 45 minutes and will include diaphragmatic breathing, systematic muscle contraction and relaxation following Jacobson's technique, controlled breathing exercises, and a brief cooldown period. The intervention will be administered by a trained physiotherapist in a group setting.
Behavioral: Functional Strength Training — Functional strength training will be delivered in weekly supervised sessions over a 10-week period. Sessions will last approximately 45 minutes and will focus on improving upper limb, lower limb, and core muscle strength using progressive resistance exercises. Training intensity will be gradually increased according to participant tolerance and performance. All sessions will be supervised by a trained physiotherapist.
  Arms: Strength Training plus Progressive Muscle Relaxation

SUMMARY:
Informal caregivers of people with Alzheimer's disease experience high physical and psychological burden, increasing their risk of frailty, anxiety, and caregiver burnout. This randomized controlled trial aims to evaluate the effectiveness of a combined strength training and progressive muscle relaxation program compared with progressive muscle relaxation alone. The intervention will last 10 weeks, with assessments conducted at baseline, post-intervention, and at a 3-month follow-up. Primary outcomes include frailty, anxiety, and caregiver burden.

DETAILED DESCRIPTION:
Alzheimer's disease is associated with long-term caregiving demands that expose informal caregivers to sustained physical and psychological stress. This chronic exposure may contribute to functional decline, increased vulnerability to frailty, and reduced overall well-being, highlighting the need for accessible, non-pharmacological interventions targeting caregiver health.

The present study adopts a parallel-group randomized controlled design in which participants are allocated to one of two intervention arms. One group will participate in structured progressive muscle relaxation sessions, while the other will receive a combined intervention integrating functional strength training with progressive muscle relaxation. The intervention protocol has been designed to be feasible, low-cost, and easily implementable in community and clinical settings.

Assessments will be conducted at multiple time points to examine changes in physical performance and psychological status over time. Standardized performance-based measures and validated self-report instruments will be used to capture functional and psychosocial outcomes, allowing for a comprehensive evaluation of the intervention effects across short- and medium-term follow-up periods.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Informal caregivers of a person with Alzheimer's disease
* Providing regular care for at least 10 hours per week
* Ability to attend intervention sessions
* Ability to understand and follow instructions
* Provision of written informed consent

Exclusion Criteria:

* Acute illness or medical conditions contraindicating participation in strength exercise
* Participation in structured exercise programs that may interfere with study outcomes
* Severe or uncontrolled psychiatric disorders
* Physical limitations preventing completion of functional assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Frailty | Baseline, 3-month follow-up and immediately after completion of the intervention (at 10 weeks).
  Frailty will be assessed using the Short Physical Performance Battery (SPPB) and handgrip strength measured with a hand dynamometer.
  The SPPB includes balance, gait speed, and lower-limb strength components. The score is obtained by summing the results of three performance-based tests: balance, gait speed over 4 meters, and the five-times sit-to-stand chair test. The total score ranges from 0 to 12 points, where 0 represents the worst performance and 12 the best performance. Lower scores (generally <10) indicate frailty and increased risk of falls. Performance is classified as follows: 0-3 (disabled), 4-6 (frail), 7-9 (prefrail), and 10-12 (independent).
  Handgrip strength will be measured using a hand dynamometer, and the absolute grip strength value will be recorded. The Fried frailty phenotype includes handgrip strength (dynamometry) as one of the five key criteria for identifying frailty in older adults. Cut-off values indicative of muscle weakness, adjusted for sex and body mass

SECONDARY OUTCOMES:
Anxiety | Baseline, 3-month follow-up and immediately after completion of the intervention (at 10 weeks)
  Anxiety symptoms will be assessed using the Hamilton Anxiety Rating Scale (HAM-A), a validated clinician-rated questionnaire evaluating psychological and somatic anxiety symptoms. HAM-A is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Caregiver burden | Baseline, 3-month follow-up and immediately after completion of the intervention (at 10 weeks)
  Caregiver burden will be assessed using the Zarit Burden Interview (ZBI), a validated self-report questionnaire measuring perceived burden in informal caregivers. The total score is calculated as the sum of all items, with a possible range from 22 to 110. Each item is rated using a 5-point Likert-type scale, with response options ranging from "never" to "almost always", scored from 1 to 5.

OTHER OUTCOMES:
Adherence to the intervention | Throughout the 10-week intervention period
  Adherence will be assessed by recording the number of sessions attended and the percentage of completed sessions for each participant.
Adverse events | Throughout the 10-week intervention period
  Adverse events or incidents occurring during the intervention sessions, such as musculoskeletal discomfort, dizziness, or other exercise-related events, will be recorded and monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will not be shared outside the study team due to ethical, privacy, and data protection considerations.